CLINICAL TRIAL: NCT02764736
Title: Atorvastatin Reduces Chronic Inflammation and aVerage Epogen Dose (ARChIVED)
Acronym: ARChIVED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment did not progress as anticipated. No participants enrolled.
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Pradhum Ram, Principal investigator, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4802
Record Dates: First submitted 2016-03-18; First posted 2016-05-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Complication of Renal Dialysis
MeSH Terms: interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atorvastatin (Experimental): Patients in this arm will receive 20mg atorvastatin PO daily for 12 weeks followed by 40mg atorvastatin PO daily for 12 weeks.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Patients will be given 20mg atorvastatin daily for 12 weeks and then increased to 40mg atorvastatin daily for an additional 12 weeks.
  Other Names: Statin

SUMMARY:
The specific aim of this trial is to determine whether initiating moderate- or high-intensity atorvastatin therapy in hemodialysis patient not previously on a statin reduces inflammation and lowers average Epogen utilization. Statin naive patients on maintenance HD will be started on 20mg atorvastatin daily for weeks and then titrated up to 40mg atorvastatin daily for an additional 12 weeks. Patient's inflammatory markers (ferritin, CRP) and weekly Epogen usage will be monitored.

DETAILED DESCRIPTION:
Patients will be identified and consented. After informed consent is obtained, baseline demographic information, past medical history, dialysis specific information, and laboratory metrics (lipid profile, inflammatory markers) will be obtained from the electronic medical records. For the first 12 weeks, all subjects will be instructed to take one 20mg atorvastatin tablet daily; atorvastatin tablets will be dispensed by the research team in 30-tablet increments every month to ensure compliance and prevent diversion. Subjects will undergo standard-of-care hemodialysis with routine hemoglobin monitoring and Epogen titration according to the dialysis center protocol. Every two weeks, they will be assessed by a research coordinator who will monitor for medication adverse effects (see attached patient survey) and medication compliance (pill counts) at alternating visits. After 12 weeks, lipid profile and inflammatory markers will be rechecked or obtained from the electronic medical record. For the subsequent 12 weeks (ie. weeks 12-24), subjects will be instructed to take two 20mg atorvastatin tablets (40mg total) daily. If the subject is unable to tolerate 40mg of atorvastatin daily due to medication adverse effects, they will continue to take 20mg atorvastatin daily for the remainder of the trial. Epogen will be titrated and subjects will be monitored as above. At the completion of the study, a lipid panel and inflammatory markers will be checked for a third time. Epogen usage and dialysis specific information will be recorded continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Stable on Hemoglobin levels on Epogen therapy (Hgb between 9.5-11.5 for prior 3 weeks)
* No statin usage during the prior 3 months
* Complaint with hemodialysis and medications

Exclusion Criteria:

* Prior history of myocardial infarction, stroke or vascular disease
* Prior hospitalization within the past 15 days
* Prior episodes of significant bleeding (trauma, GI bleed, GU bleed, menorrhagia) in the prior 15 days
* Liver disease
* Active malignancy
* Hematologic disorder

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Epoetin alfa (Epogen) utilization measured in units per week | 24 weeks
  The amount of epoetin alfa, measured in units, needed to maintain a patient's hemoglobin between 11.0 and 12.0 gm/dL

SECONDARY OUTCOMES:
C-reactive protein, ferritin levels | 24 weeks
Total cholesterol level, LDL level, HDL level | 24 weeks

IPD SHARING:
Plan to Share IPD: No